CLINICAL TRIAL: NCT04751487
Title: Randomized, Double-blind, Placebo-controlled, Parallel-group Phase 3 Study to Evaluate the Efficacy, Safety, and Tolerability of SAR440340/ REGN3500/ Itepekimab (Anti-IL-33 mAb) in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study to Assess the Efficacy, Safety, and Tolerability of SAR440340/REGN3500/Itepekimab in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: AERIFY-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC16819; U1111-1250-2843 (Registry Identifier: ICTRP); 2024-512012-21 (Registry Identifier: CTIS); 2020-001819-24 (EudraCT Number)
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — itepekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Itepekimab Q2W in former smokers (Experimental): Subcutaneous (SC) administration of Itepekimab every 2 weeks (Q2W) for up to 52 weeks
  Interventions: Drug: Itepekimab SAR440340
- Itepekimab Q4W in former smokers (Experimental): SC administration of Itepekimab every 4 weeks (Q4W) for up to 52 weeks, with alternating SC administration of matching placebo at the 2-week interval between active IMP
  Interventions: Drug: Itepekimab SAR440340; Drug: Placebo
- Placebo in former smokers (Placebo Comparator): SC administration of matching placebo Q2W for up to 52 weeks
  Interventions: Drug: Placebo
- Itepekimab Q2W in current smokers (Experimental): SC administration of Itepekimab every 2 weeks (Q2W) for 52 weeks
  Interventions: Drug: Itepekimab SAR440340
- Placebo in current smokers (Placebo Comparator): SC administration of matching placebo Q2W for 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Itepekimab SAR440340 — Pharmaceutical form: solution for injection in pre-filled syringe Route of administration: subcutaneous
  Other Names: REGN3500
  Arms: Itepekimab Q2W in current smokers; Itepekimab Q2W in former smokers; Itepekimab Q4W in former smokers
Drug: Placebo — Pharmaceutical form: solution for injection in pre-filled syringe Route of administration: subcutaneous
  Arms: Itepekimab Q4W in former smokers; Placebo in current smokers; Placebo in former smokers

SUMMARY:
Primary Objective:

Primary population (former smokers cohort):

* Evaluate the efficacy of itepekimab compared with placebo on the annualized rate of acute moderate-or-severe COPD exacerbations in former smokers with moderate-to-severe COPD

Secondary Objectives:

Primary population (former smokers cohort):

* Evaluate the efficacy of itepekimab compared with placebo on pulmonary function in former smokers with moderate-to-severe COPD
* Evaluate the efficacy of itepekimab compared with placebo on occurrence of acute exacerbation of COPD (AECOPD) in former smokers with moderate-to-severe COPD
* Evaluate the efficacy of itepekimab compared with placebo on severe AECOPD in former smokers with moderate-to-severe COPD
* Evaluate the efficacy of itepekimab compared with placebo on corticosteroid-treated AECOPD in former smokers with moderate-to-severe COPD
* Evaluate the efficacy of itepekimab compared with placebo on respiratory symptoms in former smokers with moderate-to-severe COPD
* Evaluate the efficacy of itepekimab compared with placebo on Forced Expiratory Volume in 1 second (FEV1) slope in former smokers with moderate-to-severe COPD
* Evaluate the efficacy of itepekimab compared with placebo on health-related quality of life (HRQoL) as assessed by St. George's Respiratory Questionnaire (SGRQ) in former smokers with moderate-to-severe COPD
* Evaluate the safety and tolerability of itepekimab in former smokers with moderate-to-severe COPD
* Evaluate the pharmacokinetic (PK) profile of itepekimab in former smokers with moderate-to-severe COPD
* Evaluate immunogenicity to itepekimab in former smokers with moderate-to-severe COPD

Secondary population (current smokers cohort)

* Estimate the efficacy of itepekimab compared with placebo on the annualized rate of acute moderate or severe COPD exacerbations in current smokers with moderate-to-severe COPD
* Estimate the efficacy of itepekimab compared with placebo on pulmonary function in current smokers with moderate-to-severe COPD
* Estimate the safety and tolerability of itepekimab in current smokers with moderate-to-severe COPD
* Estimate the PK profile of itepekimab in current smokers with moderate to severe COPD
* Estimate immunogenicity to itepekimab in current smokers with moderate-to-severe COPD

DETAILED DESCRIPTION:
The study duration per participant:

* Screening period is 3-5 weeks
* Randomized investigational medicinal product (IMP) treatment period is 52 weeks for first cohort of randomized former smoker participants [approximately 930] and cohort of current smokers [approximately 280], and 24 to 52 weeks for potential additional randomized former smoker participants
* Post-IMP treatment follow-up period is 20 weeks for participants not transitioning to the extension study LTS18133 Note: A long-term, double-blinded extension study (LTS18133) will be implemented to allow participants in this study to continue receiving active IMP for an additional period. Only participants completing their End-of-Treatment (EOT) visit per this study protocol will be offered to participate in the LTS18133 study.

ELIGIBILITY:
Inclusion criteria :

* Participant must be 40 to 85 years of age inclusive.
* Physician diagnosis of COPD for at least 1 year (based on Global Initiative for Chronic Obstructive Lung Disease [GOLD] definition).
* Smoking history of ≥10 pack-years:

  * For former smokers: participants who report that they are not currently smoking and smoking cessation must have occurred ≥6 months prior to Screening (Visit 1A) with an intention to quit permanently.
  * For current smokers: participants who report that they are currently smoking tobacco (participant smoked at least 1 cigarette per day on average during the past 7 days) at Screening (Visit 1A) and who are not currently participating in or planning to initiate a smoking cessation intervention at Screening (Visit 1A) or during Screening period.
* Participants with moderate-to-severe COPD
* Participant-reported history of signs and symptoms of chronic bronchitis (chronic productive cough for at least 3 months in the year prior to Screening in a participant in whom other causes of chronic cough [eg, inadequately treated gastroesophageal reflux or chronic rhinosinusitis; or clinical diagnosis of bronchiectasis] has been excluded).
* Documented history of high exacerbation risk defined as having had ≥2 moderate or ≥1 severe exacerbations within the year prior to Screening (Visit 1A), with at least 1 exacerbation treated with systemic corticosteroids. At least one exacerbation must have occurred while participants were on their current controller therapy:

  * Moderate exacerbations will be recorded by the Investigator and are defined as acute worsening of respiratory symptoms that requires either systemic corticosteroids (IM, IV, or oral) and/or antibiotics.
  * Severe exacerbations will be recorded by the Investigator and are defined as AECOPD that require hospitalization or observation for >24 hours in emergency department/urgent care facility.
* Participants with standard of care controller therapy, for ≥3 months prior to Screening (Visit 1A) and at a stable dose of controller therapy for at least 1 month prior to the Screening, including either: inhaled corticosteroid (ICS) + long-acting beta-agonist (LABA), long-acting muscarinic antagonist (LAMA) + LABA or LAMA + LABA + ICS.
* Body mass index (BMI) ≥18.0 kg/m^2, or BMI ≥16.0 kg/m^2 for participants enrolled in East-Asian countries.
* Female participant is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * not a women of child-bearing potential (WOCBP) OR
  * a WOCBP who agrees to follow the contraceptive guidance during the intervention period and for at least 20 weeks after the last dose of study intervention. -

Exclusion criteria:

* Current diagnosis of asthma according to the Global Initiative for Asthma (GINA) guidelines, or documented history of asthma unless asthma resolved before 18 years of age and has not recurred.
* For former smokers: Active smoking or vaping of any products (eg, nicotine, tetrahydrocannabinol [THC]) within 6 months prior to Screening (Visit 1A).
* For current smokers: vaping of any products (eg, nicotine, THC) within 6 months prior to Screening (Visit 1A).
* Clinically significant new abnormal electrocardiogram (ECG) within 6 months prior to, or at Screening (Visit 1A) that may affect the participant's participation in the study.
* Clinically significant and current pulmonary disease other than COPD, eg, sarcoidosis, interstitial lung disease, bronchiectasis (clinical diagnosis), diagnosis of α-1 anti-trypsin deficiency, or another diagnosed pulmonary disease.
* Diagnosis of cor pulmonale, evidence of right cardiac failure, or moderate-to-severe pulmonary hypertension.
* Hypercapnia requiring bilevel positive airway pressure (BiPAP).
* Moderate or severe exacerbation of COPD (AECOPD) within 4 weeks prior to Screening (Visit 1A).
* Prior history of / planned: lung pneumonectomy for any reason, or lung volume reduction procedures (including bronchoscopic volume reduction) for COPD. Note: Surgical biopsy, or segmentectomy, or wedge resection, or lobectomy for other diseases would not be excluded.
* Unstable ischemic heart disease, including acute myocardial infarction within the past 1 year prior to Screening, or unstable angina in the 6 months prior to Screening (Visit 1A).
* Cardiac arrhythmias including paroxysmal (eg, intermittent) atrial fibrillation.
* Uncontrolled hypertension (ie, systolic blood pressure [BP] >180 mm Hg or diastolic BP >110 mm Hg with or without use of anti-hypertensive therapy).
* Participants with active tuberculosis (TB), latent TB, a history of incompletely treated TB, suspected extrapulmonary TB infection (TBI), or who are at high risk of contracting TB (such as close contact with individuals with active or latent TB) or received Bacillus Calmette-Guérin (BCG)-vaccination within 12 weeks prior to Screening (Visit 1A).
* History of human immunodeficiency virus (HIV) infection or positive HIV 1/2 serology at Screening (Visit 1A).
* Suspicion of, or confirmed, coronavirus disease 2019 (COVID-19) infection or in contact with known exposure to COVID-19 at Screening (Visit 1A); known history of COVID-19 infection within 4 weeks prior to Screening (Visit 1A); history of requiring mechanical ventilation or extracorporeal membrane oxygenation (ECMO) secondary to COVID-19 within 3 months prior to Screening (Visit 1A); participants who have had a COVID-19 infection prior Screening (Visit 1A) who have not yet sufficiently recovered to participate in the procedures of a clinical trial.
* Evidence of acute or chronic infection requiring systemic treatment with antibacterial, antiviral, antifungal, antiparasitic, or antiprotozoal medications within 4 weeks before Screening (Visit 1A), significant viral infections within 4 weeks before Screening (Visit 1A) that may not have been treated with antiviral treatment (eg, influenza receiving only symptomatic treatment).
* Participants with active autoimmune disease or participants using immunosuppressive therapy for autoimmune disease (eg, rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis.
* History of malignancy within 5 years before Screening (Visit 1A), except completely treated in situ carcinoma of the cervix, completely treated and resolved nonmetastatic squamous or basal cell carcinoma of the skin.
* Previous use of itepekimab.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1239 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Annualized rate of moderate or severe acute exacerbation of COPD (AECOPD) in former smokers | Baseline up to End Of Treatment (EOT) (Week 52 for initial randomized participants, 24 to 52 weeks for potential additional randomized former smoker participants)
  Annualized rate of moderate or severe acute exacerbation of COPD (AECOPD) over the placebo-controlled treatment period.

SECONDARY OUTCOMES:
Change from baseline in pre-bronchodilator (BD) forced expiratory volume in 1 second (FEV1) in former smokers | Baseline to Week 24
  FEV1 is the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Change from baseline in post-BD FEV1 in former smokers | Baseline to Week 24 and Week 52
  FEV1 is the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Change from baseline in pre-BD FEV1 in former smokers | Baseline to Week 52
  FEV1 is the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time to first moderate or severe AECOPD in former smokers | Baseline through EOT (Week 52 for initial randomized participants, 24 to 52 weeks for potential additional randomized former smoker participants)
  Time to first moderate or severe AECOPD over the placebo-controlled treatment period.
Annualized rate of severe AECOPD in former smokers | Baseline up to EOT (Week 52 for initial randomized participants, 24 to 52 weeks for potential additional randomized former smoker participants)
  Annualized rate of severe AECOPD over the placebo-controlled treatment period.
Time to first severe AECOPD in former smokers | Baseline through EOT (Week 52 for initial randomized participants, 24 to 52 weeks for potential additional randomized former smoker participants)
  Time to first severe AECOPD over the placebo-controlled treatment period.
Annualized rate of corticosteroid-treated AECOPD in former smokers | Baseline up to EOT (Week 52 for initial randomized participants, 24 to 52 weeks for potential additional randomized former smoker participants)
  Annualized rate of corticosteroid-treated AECOPD over the placebo-controlled treatment period.
Change from baseline in Evaluating Respiratory Symptoms in COPD (E-RS:COPD) total score in former smokers | Baseline to Week 24 and Week 52
  The E-RS: COPD is administered as a part of the 14-item EXACT questionnaire and is completed on a daily basis.The 11-item E-RS:COPD assesses severity of respiratory symptoms overall and severity of individual symptoms such as breathlessness, cough and sputum, and chest symptoms The total score of E-RS:COPD ranges from 0 to 40, with higher values indicating more severe respiratory symptoms.
Rate of change in post-BD FEV1 (L) from baseline (post-BD FEV1 slope) in former smokers | Baseline up to EOT (Week 52 for initial randomized participants, 24 to 52 weeks for potential additional randomized former smoker participants)
Change from baseline in St. George's Respiratory Questionnaire (SGRQ) total score in former smokers | Baseline to Week 24 and Week 52
  The SGRQ is a 50-item questionnaire designed to measure and quantify health status in adult participants with chronic airflow limitation. A global score ranges from 0 to 100. Scores by dimension are calculated for 3 domains: Symptoms, Activity and Impacts (Psycho-social) as well as a total score. A lower score indicates better quality of life.
Proportion of participants with a decrease from baseline of at least 4 points in SGRQ total score in former smokers | Baseline to Week 24 and Week 52
  The SGRQ is a 50-item questionnaire designed to measure and quantify health status in adult participants with chronic airflow limitation. A global score ranges from 0 to 100. Scores by dimension are calculated for 3 domains: Symptoms, Activity and Impacts (Psycho-social) as well as a total score. A lower score indicates better quality of life.
Incidence of treatment-emergent adverse events (TEAEs), adverse event of special interests (AESIs), serious adverse events (SAEs), and adverse events (AEs) leading to permanent treatment discontinuation in former smokers | Baseline up to End-of-Study (EOS) (Up to Week 72 for participants not transitioning to the extension study LTS18133; Up to Week 52 for participants transitioning to the extension study LTS18133)
Incidence of potentially clinically significant laboratory test, vital signs, and electrocardiogram (ECGs) abnormalities in former smokers | Baseline up to EOS (Up to Week 72 for participants not transitioning to the extension study LTS18133; Up to Week 52 for participants transitioning to the extension study LTS18133)
Functional itepekimab concentrations in serum in former smokers | Baseline up to EOS (Up to Week 72 for participants not transitioning to the extension study LTS18133; Up to Week 52 for participants transitioning to the extension study LTS18133)
Incidence of treatment-emergent anti-itepekimab antibodies responses in former smokers | Baseline up to EOS (Up to Week 72 for participants not transitioning to the extension study LTS18133; Up to Week 52 for participants transitioning to the extension study LTS18133)
Annualized rate of moderate or severe AECOPD in current smokers | Baseline up to Week 52
  Annualized rate of moderate or severe AECOPD over the placebo-controlled treatment period.
Change from baseline in pre-BD FEV1 in current smokers | Baseline up to Week 24 and Week 52
  FEV1 is the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Incidence of TEAEs, AESIs, SAEs, and AEs leading to permanent treatment discontinuation in current smokers | Baseline up to EOS (Week 72 for participants not transitioning to the extension study LTS18133; Week 52 for participants transitioning to the extension study LTS18133)
Incidence of potentially clinically significant laboratory, vital signs, and ECGs abnormalities in current smokers | Baseline up to EOS (Week 72 for participants not transitioning to the extension study LTS18133; Week 52 for participants transitioning to the extension study LTS18133)
Functional itepekimab concentrations in serum in current smokers | Baseline up to EOS (Week 72 for participants not transitioning to the extension study LTS18133; Week 52 for participants transitioning to the extension study LTS18133)
Incidence of treatment-emergent anti-itepekimab antibodies responses in current smokers | Baseline up to EOS (Week 72 for participants not transitioning to the extension study LTS18133; Week 52 for participants transitioning to the extension study LTS18133)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (297):
- United States (71):
  - Synexus Phoenix Central (Central Phoenix Medical Clinic)- Site Number : 8400333, Phoenix, Arizona
  - UCSF Fresno - Site Number : 8400030, Fresno, California
  - Palmtree Clinical Research Site Number : 8400184, Palm Springs, California
  - Allianz Research Institute Colorado Site Number : 8400061, Denver, Colorado
  - Helix Biomedics, LLC - Site Number : 8400049, Boynton Beach, Florida
  - Innovative Research of West Florida, Inc- Site Number : 8400041, Clearwater, Florida
  - Beautiful Minds Clinical Research Center Site Number : 8400352, Cutler Bay, Florida
  - Omega Research - Site Number : 8400031, DeBary, Florida
  - Sciences Connections, LLC Site Number : 8400045, Doral, Florida
  - North Florida/South Georgia Veterans Health System Site Number : 8400176, Gainesville, Florida
  - Finlay Medical Research- Site Number : 8400011, Greenacres City, Florida
  - Direct Helpers Medical Center Inc- Site Number : 8400065, Hialeah, Florida
  - Multi-Specialty Research Associates, Inc- Site Number : 8400044, Lake City, Florida
  - Advanced Pulmonary Research Institute Site Number : 8400018, Loxahatchee Groves, Florida
  - Columbus Clinical Services- Site Number : 8400054, Miami, Florida
  - Finlay Medical Research Site Number : 8400007, Miami, Florida
  - MCR Research Site Number : 8400425, Miami, Florida
  - Y and L Advance Health Care, Inc D/B/A Elite Clinical Res- Site Number : 8400009, Miami, Florida
  - My Community Research Center Site Number : 8400060, Miami, Florida
  - Phoenix Medical Research- Site Number : 8400019, Miami, Florida
  - Renstar Medical Research- Site Number : 8400015, Ocala, Florida
  - Central Florida Pulmonary Group, PA- Site Number : 8400192, Orlando, Florida
  - Heuer M.D. Research Site Number : 8400016, Orlando, Florida
  - Oviedo Medical Research Site Number : 8400026, Oviedo, Florida
  - Innovation Medical Research Center- Site Number : 8400067, Palmetto Bay, Florida
  - Pines Care Research Center LLC- Site Number : 8400056, Pembroke Pines, Florida
  - Sarasota Memorial Health Care System Clinical ResearchCenter- Site Number : 8400178, Sarasota, Florida
  - Genesis Clinical Research, LLC Site Number : 8400182, Tampa, Florida
  - Clinical Research of West Florida, Inc- Site Number : 8400008, Tampa, Florida
  - Medster Research, LLC Site Number : 8400051, Valdosta, Georgia
  - North Georgia Clinical Research Site Number : 8400013, Woodstock, Georgia
  - Care Access Fairview Heights Site Number : 8400033, Fairview Heights, Illinois
  - Captain James A. Lovell Federal Health Care Center Site Number : 8400032, North Chicago, Illinois
  - Illinois Lung Institute- Site Number : 8400024, Peoria, Illinois
  - The Iowa Clinic Site Number : 8400034, West Des Moines, Iowa
  - Cotton O'Neil Garfield- Site Number : 8400063, Topeka, Kansas
  - Lexington VA Health Care System- Site Number : 8400036, Lexington, Kentucky
  - Pulmonary & Critical Care Site Number : 8400047, Shreveport, Louisiana
  - Johns Hopkins Asthma and Allergy Center- Site Number : 8400055, Baltimore, Maryland
  - Care Access Site Number : 8400276, Boston, Massachusetts
  - Care Access Site Number : 8400281, Boston, Massachusetts
  - Henry Ford Hospital Site Number : 8400052, Detroit, Michigan
  - Revive Research Institute Site Number : 8400186, Lathrup Village, Michigan
  - Washington University School of Medicine- Site Number : 8400035, St Louis, Missouri
  - Sierra Clinical Research- Site Number : 8400005, Las Vegas, Nevada
  - Smart Medical Research Site Number : 8400191, Brooklyn, New York
  - VA Western New York Healthcare System Site Number : 8400050, Buffalo, New York
  - New York - Presbyterian Queens- Site Number : 8400028, Flushing, New York
  - Schenectady Pulmonary and Critical Care Associates- Site Number : 8400029, Schenectady, New York
  - American Health Research- Site Number : 8400002, Charlotte, North Carolina
  - Advanced Respiratory and Sleep Medicine- Site Number : 8400022, Huntersville, North Carolina
  - University of Cincinnati- Site Number : 8400042, Cincinnati, Ohio
  - Remington-Davis Inc- Site Number : 8400004, Columbus, Ohio
  - Toledo Institute of Clinical Research- Site Number : 8400014, Toledo, Ohio
  - OK Clinical Research LLC- Site Number : 8400001, Edmond, Oklahoma
  - Kaiser Permanente Center for Health Research Site Number : 8400039, Portland, Oregon
  - St. Luke's University Health Network- Site Number : 8400187, Bethlehem, Pennsylvania
  - Temple University Hospital Site Number : 8400062, Philadelphia, Pennsylvania
  - Allegheny Health Network- Site Number : 8400058, Pittsburgh, Pennsylvania
  - Lowcountry Lung & Critical Care- Site Number : 8400175, Charleston, South Carolina
  - Medtrial, LLC Site Number : 8400048, Columbia, South Carolina
  - VitaLink Research- Gaffney- Site Number : 8400003, Gaffney, South Carolina
  - Clinical Trials Center of Middle Tennessee Site Number : 8400025, Franklin, Tennessee
  - TTS Research- Site Number : 8400012, Boerne, Texas
  - United Memorial Medical Center (UMMC)- Site Number : 8400193, Houston, Texas
  - Radiance Clinical Research- Site Number : 8400037, Lampasas, Texas
  - Clincove: Plano Primary Care Clinic Site Number : 8400424, Plano, Texas
  - Sun Research Institute - Site Number : 8400183, San Antonio, Texas
  - AES Salt Lake City- Site Number : 8400332, Murray, Utah
  - The Rheumatology and Pulmonary Clinic- Site Number : 8400053, Beckley, West Virginia
  - Aurora BayCare Medical Center Site Number : 8400046, Green Bay, Wisconsin
- Argentina (9):
  - Investigational Site Number : 0320009, Berazategui, Buenos Aires
  - Investigational Site Number : 0320008, CABA, Buenos Aires
  - Investigational Site Number : 0320001, CABA, Buenos Aires
  - Investigational Site Number : 0320005, Pergamino, Buenos Aires
  - Investigational Site Number : 0320006, Buenos Aires, Buenos Aires F.D.
  - Investigational Site Number : 0320002, Vicente Lopez, Buenos Aires F.D.
  - Investigational Site Number : 0320007, Rosario, Santa Fe Province
  - Investigational Site Number : 0320003, Rosario, Santa Fe Province
  - Investigational Site Number : 0320004, Rosario, Santa Fe Province
- Brazil (17):
  - CEDOES - Centro de Diagnostico e Pesquisa de Osteoporose do ES- Site Number : 0760009, Vitória, Espírito Santo
  - SER da Bahia- Site Number : 0760020, Salvador, Estado de Bahia
  - CECAP - Centro de Cardiologia Clinica e Pesquisa Dra. Juliana Souza- Site Number : 0760018, Brasília, Federal District
  - Hospital Sao Domingos- Site Number : 0760016, São Luís, Maranhão
  - Santa Casa de Belo Horizonte - Hospital Emygdio Germano- Site Number : 0760014, Belo Horizonte, Minas Gerais
  - CETI - Centro de Estudos em Terapias Inovadoras- Site Number : 0760012, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericordia de Porto Alegre- Site Number : 0760001, Porto Alegre, Rio Grande do Sul
  - Instituto Ceos Site Number : 0760021, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS- Site Number : 0760007, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao - Grupo Hospitalar Conceicao- Site Number : 0760006, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina da Universidade Estadual Paulista- Site Number : 0760005, Botucatu, São Paulo
  - PUC Campinas - Sociedade Campineira de Educaçao e Instruçao- Site Number : 0760010, Campinas, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clinicos- Site Number : 0760015, São Bernardo do Campo, São Paulo
  - Nucleo de Pesquisa Clinica e Ensino da Rede Sao Camilo- Site Number : 0760013, São Paulo, São Paulo
  - Clinica de Alergia Martti Antila Site Number : 0760008, Sorocaba, São Paulo
  - Instituto Brasil de Pesquisa Clínica-IBPCLIN S/A Site Number : 0760017, Rio de Janeiro
  - CEPIC - Centro Paulista de Investigação Clínica- Site Number : 0760004, São Paulo
- Bulgaria (10):
  - Investigational Site Number : 1000008, Blagoevgrad
  - Investigational Site Number : 1000013, Dupnitsa
  - Investigational Site Number : 1000004, Gabrovo
  - Investigational Site Number : 1000009, Haskovo
  - Investigational Site Number : 1000005, Montana
  - Investigational Site Number : 1000002, Plovdiv
  - Investigational Site Number : 1000012, Rousse
  - Investigational Site Number : 1000003, Rousse
  - Investigational Site Number : 1000001, Sofia
  - Investigational Site Number : 1000006, Sofia
- Canada (16):
  - Investigational Site Number : 1240006, Sherwood Park, Alberta
  - Investigational Site Number : 1240014, Kelowna, British Columbia
  - Investigational Site Number : 1240016, Penticton, British Columbia
  - Investigational Site Number : 1240012, Moncton, New Brunswick
  - Investigational Site Number : 1240021, Ajax, Ontario
  - Investigational Site Number : 1240020, Burlington, Ontario
  - Investigational Site Number : 1240023, Guelph, Ontario
  - Investigational Site Number : 1240009, Toronto, Ontario
  - Investigational Site Number : 1240022, Windsor, Ontario
  - Investigational Site Number : 1240018, Windsor, Ontario
  - Investigational Site Number : 1240004, Sherbrooke, Quebec
  - Investigational Site Number : 1240005, St-charles Borrommee, Quebec
  - Investigational Site Number : 1240019, Terrebonne, Quebec
  - Investigational Site Number : 1240001, Trois-Rivières, Quebec
  - Investigational Site Number : 1240002, Victoriaville, Quebec
  - Investigational Site Number : 1240003, Québec
- Chile (8):
  - Investigational Site Number : 1520009, Valdivia, Los Ríos Region
  - Investigational Site Number : 1520002, Talca, Maule Region
  - Investigational Site Number : 1520007, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520008, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Quillota, Región de Valparaíso
- Czechia (8):
  - Investigational Site Number : 2030001, Jindrichuv Hradec III
  - Investigational Site Number : 2030009, Měšice
  - Investigational Site Number : 2030005, Mladá Boleslav
  - Investigational Site Number : 2030008, Olomouc
  - Investigational Site Number : 2030004, Ostrava
  - Investigational Site Number : 2030002, Prague
  - Investigational Site Number : 2030006, Teplice
  - Investigational Site Number : 2030007, Varnsdorf
- Denmark (2):
  - Investigational Site Number : 2080001, Hvidovre
  - Investigational Site Number : 2080003, Vejle
- Investigational Site Number : 2330001, Tartu, Estonia
- France (4):
  - Investigational Site Number : 2500001, Lyon
  - Investigational Site Number : 2500002, Montpellier
  - Investigational Site Number : 2500003, Pessac
  - Investigational Site Number : 2500004, Reims
- Georgia (3):
  - Investigational Site Number : 2680003, Batumi
  - Investigational Site Number : 2680001, Tbilisi
  - Investigational Site Number : 2680002, Tbilisi
- Germany (13):
  - Investigational Site Number : 2760006, Bendorf
  - Investigational Site Number : 2760004, Berlin
  - Investigational Site Number : 2760009, Berlin
  - Investigational Site Number : 2760010, Berlin
  - Investigational Site Number : 2760005, Frankfurt am Main
  - Investigational Site Number : 2760002, Hamburg
  - Investigational Site Number : 2760014, Hanover
  - Investigational Site Number : 2760008, Leipzig
  - Investigational Site Number : 2760007, Leipzig
  - Investigational Site Number : 2760003, Lübeck
  - Investigational Site Number : 2760001, Mainz
  - Investigational Site Number : 2760012, Neu-Isenburg
  - Investigational Site Number : 2760011, Rosenheim
- Hungary (7):
  - Investigational Site Number : 3480002, Balassagyarmat
  - Investigational Site Number : 3480009, Budapest
  - Investigational Site Number : 3480005, Edelény
  - Investigational Site Number : 3480004, Hajdunánás
  - Investigational Site Number : 3480003, Püspökladány
  - Investigational Site Number : 3480001, Százhalombatta
  - Investigational Site Number : 3480012, Szombathely
- India (11):
  - Investigational Site Number : 3560016, Belagavi
  - Investigational Site Number : 3560001, Chandigarh
  - Investigational Site Number : 3560014, India
  - Investigational Site Number : 3560013, Jaipur
  - Investigational Site Number : 3560019, Kanpur
  - Investigational Site Number : 3560010, Kolkata
  - Investigational Site Number : 3560017, Nagpur
  - Investigational Site Number : 3560005, Nagpur
  - Investigational Site Number : 3560009, Nashik
  - Investigational Site Number : 3560012, Pune
  - Investigational Site Number : 3560018, Pune
- Israel (5):
  - Investigational Site Number : 3760003, Jerusalem
  - Investigational Site Number : 3760002, Jerusalem
  - Investigational Site Number : 3760001, Petah Tikva
  - Investigational Site Number : 3760009, Ramat Gan
  - Investigational Site Number : 3760004, Rehovot
- Japan (31):
  - Investigational Site Number : 3920023, Nagoya, Aichi-ken
  - Investigational Site Number : 3920020, Nagoya, Aichi-ken
  - Investigational Site Number : 3920005, Fukuoka, Fukuoka
  - Investigational Site Number : 3920027, Fukuoka, Fukuoka
  - Investigational Site Number : 3920030, Kurume-shi, Fukuoka
  - Investigational Site Number : 3920015, Mizunami-shi, Gifu
  - Investigational Site Number : 3920010, Hiroshima, Hiroshima
  - Investigational Site Number : 3920021, Kure-shi, Hiroshima
  - Investigational Site Number : 3920035, Kure-shi, Hiroshima
  - Investigational Site Number : 3920038, Sapporo, Hokkaido
  - Investigational Site Number : 3920042, Sapporo, Hokkaido
  - Investigational Site Number : 3920013, Himeji-shi, Hyōgo
  - Investigational Site Number : 3920009, Sakaide-shi, Kagawa-ken
  - Investigational Site Number : 3920014, Takamatsu, Kagawa-ken
  - Investigational Site Number : 3920011, Konan-ku, Yokohama-shi, Kanagawa
  - Investigational Site Number : 3920039, Yokohama, Kanagawa
  - Investigational Site Number : 3920043, Matsusaka-shi, Mie-ken
  - Investigational Site Number : 3920003, Osaka, Osaka
  - Investigational Site Number : 3920026, Osaka, Osaka
  - Investigational Site Number : 3920007, Sakai-shi, Osaka
  - Investigational Site Number : 3920006, Yao-shi, Osaka
  - Investigational Site Number : 3920036, Sano-shi, Tochigi
  - Investigational Site Number : 3920040, Chuo-ku, Tokyo
  - Investigational Site Number : 3920017, Chuo-ku, Tokyo
  - Investigational Site Number : 3920024, Chuo-ku, Tokyo
  - Investigational Site Number : 3920019, Itabashi-ku, Tokyo
  - Investigational Site Number : 3920029, Kiyose, Tokyo
  - Investigational Site Number : 3920025, Shibuya-ku, Tokyo
  - Investigational Site Number : 3920016, Shinagawa-ku, Tokyo
  - Investigational Site Number : 3920037, Shinagawa-ku, Tokyo
  - Investigational Site Number : 3920041, Toshima-ku, Tokyo
- Latvia (2):
  - Investigational Site Number : 4280002, Daugavpils
  - Investigational Site Number : 4280001, Riga
- Lithuania (3):
  - Investigational Site Number : 4400002, Kaunas
  - Investigational Site Number : 4400001, Kaunas
  - Investigational Site Number : 4400003, Klaipėda
- Mexico (10):
  - Investigational Site Number : 4840008, Monterrey, Nuevo León
  - Investigational Site Number : 4840009, Monterrey, Nuevo León
  - Investigational Site Number : 4840002, Monterrey, Nuevo León
  - Investigational Site Number : 4840010, Aguascalientes
  - Investigational Site Number : 4840003, Chihuahua City
  - Investigational Site Number : 4840007, Durango
  - Investigational Site Number : 4840012, Durango, Durango
  - Investigational Site Number : 4840006, Mexico City
  - Investigational Site Number : 4840001, Monterrey, Nuevo León
  - Investigational Site Number : 4840004, Veracruz
- Netherlands (3):
  - Investigational Site Number : 5280005, Arnhem
  - Investigational Site Number : 5280001, Breda
  - Investigational Site Number : 5280008, Zutphen
- Investigational Site Number : 5780001, Lørenskog, Norway
- Poland (5):
  - Investigational Site Number : 6160005, Wołomin, Masovian Voivodeship
  - Investigational Site Number : 6160008, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160003, Malbork, Pomeranian Voivodeship
  - Investigational Site Number : 6160002, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160009, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Portugal (5):
  - Investigational Site Number : 6200009, Almada
  - Investigational Site Number : 6200006, Aveiro
  - Investigational Site Number : 6200002, Braga
  - Investigational Site Number : 6200001, Guimarães
  - Investigational Site Number : 6200010, Matosinhos Municipality
- Puerto Rico (4):
  - Cardiopulmonary Research- Site Number : 8400040, Guaynabo
  - BRCR Medical Center, Inc. Site Number : 8400190, Ponce
  - BRCR Medical Center Site Number : 8400180, San Juan
  - Inspire Pulmonary & Sleep Medicine Specialists Site Number : 8400232, Temecula
- Russia (6):
  - Investigational Site Number : 6430002, Moscow
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430005, Moscow
  - Investigational Site Number : 6430004, Saint Petersburg
  - Investigational Site Number : 6430003, Saint Petersburg
  - Investigational Site Number : 6430006, Ulyanovsk
- South Africa (12):
  - Investigational Site Number : 7100013, Benoni
  - Investigational Site Number : 7100019, Cape Town
  - Investigational Site Number : 7100002, Cape Town
  - Investigational Site Number : 7100015, Chatsworth
  - Investigational Site Number : 7100005, Durban
  - Investigational Site Number : 7100017, Durban
  - Investigational Site Number : 7100006, Durban
  - Investigational Site Number : 7100016, Durban
  - Investigational Site Number : 7100004, Gatesville
  - Investigational Site Number : 7100012, Middelburg
  - Investigational Site Number : 7100003, Parow
  - Investigational Site Number : 7100009, Pretoria
- South Korea (5):
  - Investigational Site Number : 4100002, Wŏnju, Gangwon-do
  - Investigational Site Number : 4100005, Seongnam-si, Gyeonggi-do
  - Investigational Site Number : 4100003, Incheon, Incheon-gwangyeoksi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul
- Spain (12):
  - Investigational Site Number : 7240004, Palma de Mallorca, Balears [Baleares]
  - Investigational Site Number : 7240014, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240006, Sant Boi de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240013, Santander, Cantabria
  - Investigational Site Number : 7240002, Mérida / Badajoz, Extremadura
  - Investigational Site Number : 7240009, Lleida / Lleida, Lleida [Lérida]
  - Investigational Site Number : 7240008, Pozuelo de Alarcón, Madrid
  - Investigational Site Number : 7240007, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240010, Cáceres
  - Investigational Site Number : 7240003, Madrid
  - Investigational Site Number : 7240001, Málaga
  - Investigational Site Number : 7240012, Zaragoza
- Turkey (Türkiye) (6):
  - Investigational Site Number : 7920007, Ankara
  - Investigational Site Number : 7920005, Balcali Adana
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920003, Izmir
  - Investigational Site Number : 7920006, Kırıkkale
  - Investigational Site Number : 7920002, Mersin
- United Kingdom (7):
  - Investigational Site Number : 8260006, Wishaw, Glasgow City
  - Investigational Site Number : 8260007, Tyne and Wear, North Tyneside
  - Investigational Site Number : 8260002, Chertsey, Surrey
  - Investigational Site Number : 8260003, Bradford
  - Investigational Site Number : 8260005, Liverpool
  - Investigational Site Number : 8260008, Milton Keynes
  - Investigational Site Number : 8260001, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC16819 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25255&tenant=MT_SNY_9011